CLINICAL TRIAL: NCT07244861
Title: Acute Effects of Transcutaneous Electrical Nerve Stimulation on Passive Muscle Stiffness and Pain in Patients With Neck Pain: A Randomized Controlled Trial
Brief Title: Acute Effects of TENS on Cervical Muscle Stiffness and Pain in Neck Pain
Acronym: TENS-NECK
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Amasya University (Other); Bangor University (Other); Ataturk University (Other)
Responsible Party: Principal Investigator, esedullah akaras, Dr., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETU-TENS-NECK-RCT-02; Erzurum Technical University (Other: Erzurum Technical University)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Neck Pain; Chronic Neck Pain; Muscle Stiffness; Transcutaneous Electrical Nerve Stimulation
Keywords: TENS; MyotonPro; VAS pain
MeSH Terms: conditions — Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Two parallel arms with 1:1 allocation (TENS vs control/sham). Randomization is computer-generated with allocation concealment using sequentially numbered, opaque, sealed envelopes (SNOSE). Outcomes are assessed pre-session and immediately post-session in a single visit. Outcome assessors are blinded; participant blinding is applied if the sham TENS arm is used.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation. Participants are not blinded when the comparator is "no intervention." If a sham TENS comparator is used, participants will also be blinded (double-blind: participant and outcomes assessor). Randomization is concealed using sequentially numbered, opaque, sealed envelopes (SNOSE); assessors do not have access to the allocation list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): Participants receive a single session of conventional TENS targeting painful/stiff cervical muscle regions (typically upper trapezius ± suboccipital) with immediate post-session assessments.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Device: Sham TENS
- Sham TENS (Sham Comparator): Participants undergo a sham stimulation session with identical setup and timing to mimic TENS without delivering therapeutic current.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Device: Sham TENS

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Conventional mode TENS, frequency ~80 Hz, pulse width ≤150 µs, duration 20 minutes. Intensity set to "strong but tolerable" without visible muscle contraction. Electrodes placed bilaterally over the most painful/stiff segments (e.g., upper trapezius midpoint along C7-acromion line; adjustments per comfort
  Other Names: Conventional TENS; TENS therapy
Device: Sham TENS — Electrodes applied at the same anatomical sites as the active arm. Device indicators remain on; intensity is ramped to perception briefly and then reduced to sub-sensory/zero so that no effective current is delivered for the remainder of the 20-minute session. Procedures and clinician-participant interactions mirror the active arm
  Other Names: Placebo TENS

SUMMARY:
This randomized controlled trial investigates the acute effects of transcutaneous electrical nerve stimulation (TENS) on passive cervical muscle stiffness (MyotonPro "dynamic stiffness", N/m) and pain (0-10 VAS) in adults with chronic/mechanical neck pain. Participants will be allocated 1:1 to TENS or control/sham. Outcomes are measured immediately before and immediately after a single 15-minute session.

DETAILED DESCRIPTION:
Background/Rationale: TENS modulates superficial afferent input and may reduce pain and muscle tone. However, its immediate impact on objective passive muscle stiffness measured by a handheld myotonometer (MyotonPro) in neck pain is insufficiently characterized. This trial tests whether a brief, low-risk intervention produces measurable changes in mechanical muscle properties and perceived pain in a short time window.

Objectives/Hypotheses:

Primary objective: Determine whether conventional TENS acutely reduces dynamic stiffness of the upper trapezius compared with control/sham.

Secondary objectives: Evaluate pain (VAS), additional MyotonPro parameters (frequency/tone, logarithmic decrement, relaxation time, creep), and safety/tolerability.

Hypothesis: TENS will show a significant group × time interaction favoring TENS over control/sham.

Design: Single-center (optionally multi-center), parallel-group, randomized (1:1) RCT. Masking: at minimum outcome assessor-blinded; participant blinding if sham TENS is used.

Sample Size: n = 24 (12 per arm), based on a priori power analysis (f≈0.40, α=0.05, power=0.95) for a 2×2 mixed design.

Intervention (TENS): Conventional mode; ~80 Hz, ≤150 µs pulse width; 15 minutes; intensity "strong but tolerable" without visible muscle contraction. Electrodes placed over the most painful/stiff segments (typically upper trapezius and/or suboccipital region), preferably bilateral.

Control/Sham: No intervention or sham TENS (electrodes applied; intensity raised to sensation then reduced below perception/zero; device indicators remain on).

Assessments & Timing:

Time points: T0 (pre-session), T1 (immediately post-session).

Primary outcome: Upper trapezius dynamic stiffness (N/m)-three repetitions averaged at a standardized anatomical landmark.

Secondary outcomes: Pain VAS (0-10); MyotonPro frequency/tone, decrement, relaxation time, creep on upper trapezius ± SCM ± cervical extensors; adverse events/tolerability. (Neck Disability Index may be collected at baseline for descriptive characterization.)

Statistical Plan: Mixed-effects repeated-measures analysis with Group (TENS vs control/sham) × Time (T0 vs T1); assumption checks with robust alternatives/transformations as needed; multiple-comparison controls; effect sizes reported.

Eligibility (summary): Adults 18-50 years with neck pain VAS ≥3/10. Key exclusions include pacemaker, pregnancy, recent invasive procedures (≤6 weeks), significant dermatologic issues at electrode sites, cervical radiculopathy/neurological signs, acute neck injury. (Full list in Eligibility.)

Safety: Low-risk, non-invasive procedure. Expected adverse effects are minor (e.g., transient discomfort or skin irritation). AE/SAE monitoring is prospective; the session will be stopped if intolerable symptoms occur.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years.

Neck pain VAS ≥ 3/10 at screening and on test day.

Clinical diagnosis of chronic or mechanical neck pain (≥6 weeks).

Able to understand study procedures and provide written informed consent.

Willing to refrain from analgesics/muscle relaxants and vigorous neck/shoulder exercise for 24 hours before testing.

Exclusion Criteria:

* Cervical radiculopathy or neurological signs (myotomal weakness, dermatomal sensory loss, reflex changes).

Recent invasive procedures to the neck/shoulder (e.g., surgery, injections, radiofrequency/neurotomy) within 6 weeks.

Pacemaker/implantable cardioverter, or other active implanted electronic device.

Pregnancy or planning pregnancy.

Skin conditions at electrode sites (open wounds, infection, severe dermatitis) or known allergy to electrode adhesive/gel.

History of epilepsy or unexplained syncope.

Acute neck trauma (<6 weeks) or red flags (fracture, malignancy, infection, inflammatory rheumatic disease).

Systemic disorders likely to affect outcomes (e.g., uncontrolled diabetes with neuropathy, severe cardiovascular disease, fibromyalgia with widespread pain).

Ongoing electrotherapy to the neck region or botulinum toxin injections to cervical muscles within 3 months.

Inability to comply with procedures (e.g., severe communication/cognitive impairment), or insufficient proficiency in Turkish to complete measures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in upper trapezius dynamic stiffness | Pre-session (T0) and immediately post-session (T1; within 5 minutes of session end)
  Passive muscle dynamic stiffness (N/m) measured with MyotonPro at a standardized landmark on the upper trapezius (midpoint along the C7-acromion line; side = most symptomatic or bilateral mean).

SECONDARY OUTCOMES:
Change in pain intensity | T0 and immediately post-session
  0-10 Visual Analog Scale for current neck pain (0 = no pain, 10 = worst imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan YAGİZ, Dr., Study Director — Amasya University
Locations (1):
- Erzurum Technical University Faculty of Health Sciences, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified IPD (outcomes, baseline demographics, allocation, adverse events) will be shared ~6 months after primary completion for 36 months via an institutional repository or encrypted transfer managed by Erzurum Technical University.